CLINICAL TRIAL: NCT04618471
Title: Study to Demonstrate the Value of Paresthesia-Free Fast-Acting Subperception (FAST) and Other SCS Therapies Using WaveWriter™ Spinal Cord Stimulator Systems in the Treatment of Chronic Pain
Brief Title: Paresthesia-Free Fast-Acting Subperception (FAST) Study
Acronym: FAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4099
Record Dates: First submitted 2020-10-31; First posted 2020-11-06 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- WaveWriter Settings (Experimental)
  Interventions: Device: Boston Scientific WaveWriter SCS System

INTERVENTIONS:
Device: Boston Scientific WaveWriter SCS System — WaveWriter SCS Programming

SUMMARY:
Study to evaluate the effectiveness of FAST-SCS (fast-acting paresthesia-free therapy) and additional SCS therapy options in patients with chronic pain using Boston Scientific WaveWriter SCS Systems.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic pain (predominantly neuropathic) of the trunk and/or limbs for at least 6 months with back pain greater or equal to leg pain.
* 22 years of age or older when written informed consent is obtained
* Able to independently read and complete all questionnaires and assessments provided in English
* Signed a valid, IRB-approved informed consent form (ICF) provided in English

Key Exclusion Criteria:

* Any pain-related diagnosis or medical/psychological condition or external factors that, in the clinician's best judgment, might confound reporting of study outcomes
* Significant cognitive impairment that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to participate in the study
* Breast-feeding or planning to get pregnant during the course of the study or not using adequate contraception
* Participating, or intends to participate, in another clinical trial that may influence the data that will be collected for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2029-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (13):
- United States (13):
  - Vitamed Research, Palm Desert, California
  - Denver Back Pain Specialists, Greenwood Village, Colorado
  - Orlando Health Neuroscience Institute, Clermont, Florida
  - The Orthopaedic Institute, Gainesville, Florida
  - University of Chicago Hospital, Chicago, Illinois
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Acute and Chronic Pain Therapies, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only consented subjects who meet protocol criteria proceed to activation. The primary endpoint analysis is based on 20 activated subjects at 3-Month Visit. At the time of analysis, 104 provided informed consent, of which 62 were screen failures, 11 were withdrawn. Of the 31 remaining subjects 9 were pending evaluation, 2 had IPG activation and 20 had completed the 3-Month Visit. 73 additional subjects were consented before enrollment was complete. This accounts for the 177 subjects (104+73).
Period: Overall Study
Arm/Group | WaveWriter Settings
Started | 177
Completed | 20
Not Completed | 157
Not completed — Screen Failure | 62
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1
Not completed — Various other reasons | 2
Not completed — Pending study evaluation and completion of 3-Month post activation visit | 84

BASELINE CHARACTERISTICS:
Population: Subjects who had completed Baseline Visit at the time of the pre-specified interim analysis of 20 activated subjects at 3-month interim visit. The data reported is from a pre-specified interim analysis.
Arm/Group | WaveWriter Settings
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.67 (13.08)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 56
  Gender: Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black, of African heritage | 13
  Race: Caucasian | 65
  Race: Hispanic or Latino | 5
  Race: Native Hawaiian or other Pacific Islander | 1
  Race: Not disclosed | 2
Region of Enrollment [Number; unit: participants]
  United States | 86
Average overall pain (VRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity is expressed on a 0 - 10 verbal rating scale (VRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine". Population: At the time of analysis, three subjects had no completed the Baseline VRS questionnaire.
  units on a scale
    number analyzed (Participants) | 83
    (all) | 7.4 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Targeted Pain Responder Rate
Description: Proportion of subjects with 50% or greater reduction from Baseline Visit in average targeted pain intensity at 3 months post-activation
Time Frame: 3 months post-activation
Population: Interim analysis of 20 activated subjects at 3-Month Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | WaveWriter Settings
Number analyzed (Participants) | 20
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse Event Rates for all Subjects at time of the pre-specified primary endpoint analysis for 20 activated subjects at 3-Month Visit, approximately 7-8 months post informed consent.
Arm/Group | WaveWriter Settings
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 6/104
Other Adverse Events (participants affected / at risk) | 6/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WaveWriter Settings (N=104)
Pneumonia (Infections and infestations) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WaveWriter Settings (N=104)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Implant site pain (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Device stimulation issue (Product Issues) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT04618471/Prot_SAP_000.pdf